CLINICAL TRIAL: NCT03589950
Title: A Parallel Control, Exploratory Trial to Compare Anlotinib Plus Chemotherapy Versus Chemotherapy as Second-line Treatment in Subjects With Advanced Non-small Cell Lung Cancer
Brief Title: Anlotinib Plus Chemotherapy for Patients With Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anlo01
Record Dates: First submitted 2018-06-22; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Lung Neoplasms; Docetaxel; Pemetrexed; S-1; Anlotinib
Keywords: anlotinib; docetaxel; pemetrexed
MeSH Terms: conditions — Lung Neoplasms | interventions — anlotinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib plus chemotherapy (Experimental): Anlotinib (12mg QD PO d1-14, 21 days per cycle) + Docetaxel (75mg/m2 IV d1)/Pemetrexed (500 mg/m2 IV d1), q21d/S-1 (80-120mg/day,depending on body surface area; days 1-28 in a 6-week cycle)
  Interventions: Drug: anlotinib plus chemotherapy
- Chemotherapy (Active Comparator): Docetaxel (75mg/m2 IV d1)/Pemetrexed (500 mg/m2 IV d1), q21d/S-1 (80-120mg/day,depending on body surface area; days 1-28 in a 6-week cycle)
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: anlotinib plus chemotherapy — Anlotinib (12mg QD PO d1-14, 21 days per cycle), Docetaxel (75mg/m2 IV d1)/Pemetrexed (500 mg/m2 IV d1), q21d/S-1 (80-120mg/day,depending on body surface area; days 1-28 in a 6-week cycle)
  Arms: Anlotinib plus chemotherapy
Drug: chemotherapy — Docetaxel (75mg/m2 IV d1)/Pemetrexed (500 mg/m2 IV d1), q21d/S-1 (80-120mg/day,depending on body surface area; days 1-28 in a 6-week cycle)
  Arms: Chemotherapy

SUMMARY:
Anlotibib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit. It has the obvious resistance to new angiogenesis. The trial is to explore Anlotinib for the effectiveness and safety of advanced non-small cell lung cancer who failed first lines of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 -2
3. Subjects with histologically or cytologically confirmed locally advanced or advanced NSCLC who have previously received one lines chemotherapy, EGFR TKI or ALK inhibitor (whom with EGFR or ALK mutation but not with T790 M positive) treatment before participating；
4. Subjects with at least one measurable lesion as defined by RECIST (version 1.1),which is confirmed by computed tomography (CT) scan or MRI .
5. Subjects without brain metastases or asymptomatic brain metastases, and not needing for dehydrating agents or corticosteroids to control intracranial symptoms;
6. Survival expectation ≥ 3 months;
7. The main organ function is normal;
8. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative.
9. Subjects provided written informed consent before participating, willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Small Cell Lung Cancer; 2. Subjects with symptomatic brain metastases; 3. Survival expectation < 3 months; 4. examined as positive in EGFR&ALK mutation detection and never take the treatment of TKIs 5. Blood transfusion is required in the first dose of drug treatment within 14 days ; 6. The interval of subjects had received chemotherapy, biotherapy, radiotherapy or other anticancer therapies in the first dose of drug treatment within 21 days(excluding palliative radiotherapy); 7. The risk of active bleeding; 8. Subjects with uncontrolled blood pressure with medication (140/90 mmHg) 9. Laboratory values and organ functions ： （1）Hematologic insufficiency:

1. Hemoglobin (Hb)<8.5 g/dL，
2. Absolute neutrophil count (ANC)≤1.5×109/L，
3. Platelet count (PLT)< 100×109/L； （2）Insufficient liver function:
4. Bilirubin > 1.5×the upper limit of normal (ULN)
5. Alanine aminotransferase (ALT), or Aspartate aminotransferase (AST) >3.0×(ULN), When liver metastases,Bilirubin > 1.5×ULN, ALT or AST >5.0×(ULN.
6. serum creatinine ≤1.0×（ULN）, or creatinine clearance > 50 mL/min( calculated per the Cockcroft and Gault formula) (3) Subjects with positive for HBV surface antigen ( HBsAg)or anti-hcv (4)Subjects with Interstitial lung disease (5)Insufficient renal function: serum creatinine≥ 1.5×（ULN）, or creatinine clearance <60 mL/min

10. impairment of heart function: (1)Left ventricular ejection fraction (LVEF) <45% (LVEF evaluation is not required for subjects have no history of congestive heart failure), (2)Unstable angina, (3)Severe arrhythmia, (4)NYHA III or IVgrade of congestive heart failure, (5) Subjects with myocardial infarction within the last 12 months before entering the trial, (6)Pericardial effusion, 11. Subjects with liver fibrosis or hepatic cirrhosis 12. (1)Subjects with other active malignancy (except for definitively treated non melanoma skin cancer,carcinoma in-situ of the cervix,or other cancers that are treated with curative treatment and have no signs of recurrence for at least 5 years ) , (2)Subjects with dysphagia,malabsorption,chronic gastrointestinal diseases,or other medical history may hinder compliance and / or experimental drug absorption, 13. Subjects with major surgery in the first dose of drug treatment within 28 days, 14. Subjects with positive unknown human immunodeficiency virus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  progression-free survival
DCR | Time Frame: each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate

SECONDARY OUTCOMES:
OS | From randomization until death (up to 24 months)
  Overall survival
ORR | each 21 days up to the toxicity or PD (up to 24 months)
  Objective Response Rate
Quality of life score | each 21 days up to the toxicity or PD (up to 24 months)
  Quality of life score
Safety | each 21 days up to the toxicity or PD (up to 24 months)
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Lianyungang Hospital of Xuzhou Medical University, Lianyungang, Jiangsu, China

REFERENCES:
- [Background] Xie C, Wan X, Quan H, Zheng M, Fu L, Li Y, Lou L. Preclinical characterization of anlotinib, a highly potent and selective vascular endothelial growth factor receptor-2 inhibitor. Cancer Sci. 2018 Apr;109(4):1207-1219. doi: 10.1111/cas.13536. Epub 2018 Mar 25. PMID 29446853
- [Background] Sun Y, Niu W, Du F, Du C, Li S, Wang J, Li L, Wang F, Hao Y, Li C, Chi Y. Safety, pharmacokinetics, and antitumor properties of anlotinib, an oral multi-target tyrosine kinase inhibitor, in patients with advanced refractory solid tumors. J Hematol Oncol. 2016 Oct 4;9(1):105. doi: 10.1186/s13045-016-0332-8. PMID 27716285
- [Background] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373